CLINICAL TRIAL: NCT03218241
Title: A Randomized, Double-Blind, Placebo-Controlled Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenously Administered PRT064445, a Factor Xa (fXa) Inhibitor Antidote
Brief Title: Single Ascending Dose Study of PRT064445, a Factor Xa (fXa) Inhibitor Antidote
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 11-501
Record Dates: First submitted 2012-12-27; First posted 2017-07-14 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — PRT064445

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- PRT0064445 Dose 1 (Experimental): Dose 1 versus Placebo
  Interventions: Biological: PRT064445; Drug: Placebo
- PRT064445 Dose 2 (Experimental): Dose 2 versus Placebo
  Interventions: Biological: PRT064445; Drug: Placebo
- PRT064445 Dose 3 (Experimental): Dose 3 versus Placebo
  Interventions: Biological: PRT064445; Drug: Placebo
- PRT064445 Dose 4 (Experimental): Dose 4 versus Placebo
  Interventions: Biological: PRT064445; Drug: Placebo
- PRT064445 Dose 5 (Experimental): Dose 5 versus Placebo
  Interventions: Biological: PRT064445; Drug: Placebo

INTERVENTIONS:
Biological: PRT064445 — Intravenous
Drug: Placebo — Intravenous to mimic PRT064445
  Other Names: Placebo (for PRT064445)

SUMMARY:
This is a single center, double-blind, randomized, placebo-controlled, ascending, single dose study of PRT064445 or its matching placebo, in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women between the ages of 18 and 50 years old, inclusive
* BMI 19-32 and weighs at least 60kgs

Exclusion Criteria:

* History or symptoms of bleeding problems or thrombotic conditions
* Clinically significant medical history
* Major surgery, severe trauma, or bone fracture within 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics assessments | Up to 28 days

SECONDARY OUTCOMES:
Pharmacokinetics: Plasma levels of PRT064445 | Up to 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Phoenix, Arizona, United States